CLINICAL TRIAL: NCT05711290
Title: In Vivo Double-blind, Randomized, Placebo Controlled, Crossover Investigation of the Effect of Oral Administration of Oxygen Nanobubbles on the Distance Covered in a 6 Minute Walk Test in Patients With Pulmonary Fibrosis
Brief Title: Oxygen Nanobubble Drink Impact on Exercise in Pulmonary Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 308993
Record Dates: First submitted 2023-01-16; First posted 2023-02-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen Nanobubble First (Experimental): In this arm, the oxygen nanobubbles will be provided as a drink first. The oxygen nanobubbles mixture will be mixed with water and oxygenated. This will be provided as a one-time 200ml drink 10 minutes before the start of the 6 minute walk test.
  In this arm, the placebo will be provided as the second drink. This will be provided after atleast 2 hours after the first 6 minute walk test is completed. The placebo mixture will be mixed with water and oxygenated. This will be provided as a one-time 200ml drink 10 minutes before the start of the 6 minute walk test.
  Interventions: Dietary Supplement: Oxygen Nanobubble; Other: Placebo
- Placebo First (Placebo Comparator): In this arm, the placebo will be provided as a drink first. The placebo mixture will be mixed with water and oxygenated. This will be provided as a one-time 200ml drink 10 minutes before the start of the 6 minute walk test.
  In this arm, the oxygen nanobubbles will be provided as the second drink. This will be provided after atleast 2 hours after the first 6 minute walk test is completed. The oxygen nanobubbles mixture will be mixed with water and oxygenated. This will be provided as a one-time 200ml drink 10 minutes before the start of the 6 minute walk test.
  Interventions: Dietary Supplement: Oxygen Nanobubble; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Oxygen Nanobubble — This intervention consists of oxygenated nanobubbles made from lecithin with natural flavourings (liquorice, glycerol and citric acid)
Other: Placebo — The placebo does not contain nanobubbles, and is made from natural flavourings (liquorice, glycerol and citric acid).

SUMMARY:
Approximately 1 in 5 (or 12.7 million adults) in the UK have longstanding respiratory illnesses, and 6.5 million patients report taking prescription medication to ease the burden. Many patients suffer from lung tissue damage, which impairs adequate blood oxygenation and reduces blood saturations, and causes breathlessness. The current method of treatment is palliative - with the patient breathing supplemental oxygen through an oxygen cylinder and tube. This severely compromises patients' quality of life, as they are tethered to a heavy, unwieldy oxygen cylinder, limiting their ability and willingness to leave home.

Several recent studies in both animals and humans have indicated that orally administered oxygenated nanobubbles is a safe intervention that can improve tissue oxygenation. This randomized, double-blinded, cross-over, placebo-controlled study will evaluate the effect of an oxygen nanobubbles drink on the exercise performance of patients with chronic lung disease, such as pulmonary fibrosis. Patients will conduct the 6 Minute Walk Test (6MWT) twice, once with a placebo drink and once with the oxygen nanobubbles drink, based on a double-blind randomization protocol, and this study will evaluate the distance walked, heart rate, oxygen levels, breathlessness, and time to recovery in both cases. The investigators hypothesize that drinking the oxygen nanobubbles drink will improve the delivery of oxygen to vital organs, improving the distance a patient can cover in the 6 Minute Walk Test by 30m, which is the minimum clinically important difference.

ELIGIBILITY:
Inclusion Criteria:

* Patient is Male or Female, aged 18 years or above
* Participant is willing and able to give informed consent for participation in the study.
* Patients diagnosed with Pulmonary Fibrosis as per ATS/ERS guidelines, and in whom the lung fibrosis is considered the dominant cause of symptoms (i.e. no severe other disease such as COPD or heart failure)
* The patient must be able to walk independently without a walking stick
* The patient can, in the view of their respiratory clinician, adequately participate in a 6MW test

Exclusion Criteria:

* Pregnant or breast feeding
* History of current neurological condition (e.g., epilepsy)
* Patient has consumed liquorice in the last 24 hours.
* Patients with TLCO <30%
* Patients with known unstable ischaemic heart disease or pulmonary hypertension
* Patients with a history of smoking in the previous 30 days
* Patients that are allergic or intolerant towards: Liquorice, Lecithin derived from soya or sunflower, Citric acid, Glycerol
* Patients with known severe Renal Dysfunction
* Patients with known severe Liver Dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Distance | 1 day
  Distance covered in 6 Minute Walk Test (6MWT) with oxygen nanobubbles drink compared with placebo drink

SECONDARY OUTCOMES:
Breathlessness | 1 day
  Changes in the Modified Borg score before and after the 6MWT with oxygen nanobubbles drink compared with placebo drink
  The Modified Borg (mBORG) scale from 0-10, with a higher score denoting less breathlessness and a better patient outcome.
Heart Rate | 1 day
  Heart Rate changes in 6MWT with oxygen nanobubbles drink compared with placebo drink
Oxygen Saturation | 1 day
  SpO2 changes in 6MWT with oxygen nanobubbles drink compared with placebo drink
Recovery Time | 1 day
  Time for SpO2 and HR to reset to resting levels after 6MWT with oxygen nanobubbles drink compared with placebo drink
Patient Perception of Exercise Ability | 1 day
  Patient self-reporting via patient questionnaire the additional distance they believe they can walk after 6MWT with oxygen nanobubbles drink compared with placebo drink

CONTACTS AND LOCATIONS:
Overall Officials: Najib Rahman, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No